CLINICAL TRIAL: NCT02740348
Title: Point-of-Care Follow-Up With Primary Care After Emergency Department Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Melissa McCarthy, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 091554
Record Dates: First submitted 2016-04-13; First posted 2016-04-15 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Conditions Influencing Health Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ZocDoc Assistance (Experimental): Research assistant sets up follow-up appointment for subject using ZocDoc.
  Interventions: Behavioral: ZocDoc Assistance
- ZocDoc Information (Active Comparator): Research assistance provides subject with written information about ZocDoc.
  Interventions: Behavioral: ZocDoc Information
- Usual Care (No Intervention): ED staff gives written and verbal discharge instructions to subject.

INTERVENTIONS:
Behavioral: ZocDoc Assistance — Research assistant sets up a follow-up appointment for a subject with a primary care doctor using ZocDoc
  Arms: ZocDoc Assistance
Behavioral: ZocDoc Information — Providing ZocDoc information to subjects so that they can make a follow-up appointment with a primary care doctor themselves
  Arms: ZocDoc Information

SUMMARY:
The purpose of this trial is to determine whether setting up a follow-up appointment for patients who received treatment and were discharged from the emergency department increases their compliance with the follow-up appointment. We are enrolling patients who need a follow-up visit, have health insurance but report do not have a primary care doctor. Patients are randomized to one of three treatment groups: (1) assistance setting up a follow-up appointment by a research assistant using ZocDoc; (2) ZocDoc information given to the subject to set up follow-up appointment by him/herself; or (3) usual discharge instructions by ED staff. Subjects are phoned approximately 2 weeks after the ED visit and asked whether they completed a follow-up visit, satisfaction with their ED visit, satisfaction with their follow-up visit, and additional ED treatment and recovery.

DETAILED DESCRIPTION:
This is a randomized controlled trial involving adult emergency department (ED) patients who need a follow-up visit as defined by the ED provider (importance of follow-up rated as 5 or greater on a 0 to 10 scale). There is software available called ZocDoc that provides a user the ability to identify primary care providers who have open appointments and will take the person's health insurance (in network and outside of network) and list the doctors based on their proximity to the person in need. We are testing whether booking appointments for ED patients using ZocDoc vs. giving patients the information to use ZocDoc themselves vs. standard discharge instructions given by ED staff (i.e. you should follow-up with a primary care doctor) affects compliance with self-reported follow-up visits. We are enrolling patients while they are in the ED, completed a short baseline interview and then another interview with them over the telephone approximately two weeks after the index ED visit. The follow-up interview asks subjects whether they have completed a follow-up visit, satisfaction with the ED visit and the primary care visit, any other additional ED treatment and extent of recovery from the problem that brought them to the ED the first time.

ELIGIBILITY:
Inclusion Criteria: Patients with health insurance but report not having a primary care provider and are rated by the ED provider as needing a follow-up visit with a primary care provider (rated as moderate to high need by ED provider).

-

Exclusion Criteria: Patients doesn't want a primary care provider or patient doesn't want a follow-up visit. Patient is unable to understand consent, is a prisoner, or does not have access to email (because ZocDoc sends appointment information to email).

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Self-reported follow-up visit | 2-4 weeks after the index ED visit
  patient-reported follow-up visit with a primary care doctor

SECONDARY OUTCOMES:
Satisfaction with the ED visit | Measured 2 weeks after the index ED visit
  patient-reported satisfaction rating
Satisfaction with the primary care visit | 2-4 weeks after the index ED visit
  patient-reported satisfaction rating
Recovery from health problem | 2-4 weeks after the index ED visit
  patient-reported resolution of problem that they reported during index ED visit
Additional ED visit(s) | 2-4 weeks after the index ED visit
  Did patient receive additional ED treatment for same problem as index ED visit

CONTACTS AND LOCATIONS:
Overall Officials: Tina Choudri, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Doran KM, Colucci AC, Hessler RA, Ngai CK, Williams ND, Wallach AB, Tanner M, Allen MH, Goldfrank LR, Wall SP. An intervention connecting low-acuity emergency department patients with primary care: effect on future primary care linkage. Ann Emerg Med. 2013 Mar;61(3):312-321.e7. doi: 10.1016/j.annemergmed.2012.10.021. Epub 2012 Dec 20. PMID 23261312
- [Background] Chan TC, Killeen JP, Castillo EM, Vilke GM, Guss DA, Feinberg R, Friedman L. Impact of an internet-based emergency department appointment system to access primary care at safety net community clinics. Ann Emerg Med. 2009 Aug;54(2):279-84. doi: 10.1016/j.annemergmed.2008.10.030. Epub 2008 Dec 13. PMID 19070939